CLINICAL TRIAL: NCT06598280
Title: Same-Day Discharge Versus Overnight Stay Following Pulmonary Vein Isolation for Atrial Fibrillation - the SHAzAM-AF Study
Brief Title: Same-Day Discharge Versus Overnight Stay Following Pulmonary Vein Isolation for Atrial Fibrillation
Acronym: SHAzAM-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Roland Richard Tilz, MD, Prof. Dr. univ. med., University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHAzAM-AF
Record Dates: First submitted 2024-07-12; First posted 2024-09-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SDD Group (Experimental): Following successful venipuncture, one or two PPS are deployed at the discretion of the operator prior to catheter insertion for catheter sheath sizes ≥ 9 French. Another PPS is deployed after catheter removal if the sheath size is < 9 French. All sheaths are removed at the end of the ablation procedure. Hemostasis should be achieved by delivery of the suture. Protamine may be administered according to institutional standards. A vertical mattress suture (Donati suture) is applied superficially to conform to the skin tissue. The suture is removed on the first day after PVI.
  Interventions: Procedure: Atrial Fibrillation with femoral closure using closing system
- ONS Group (Experimental): Once the PVI block is confirmed, a figure-of-eight suture is placed at the femoral access site. The sheaths are removed and haemostasis should be achieved by manual compression at the discretion of the operator. Protamine may be administered according to institutional standards. A tourniquet is applied for a minimum of 30 minutes and the patient should remain supine.
  Interventions: Procedure: Atrial Fibrillation with femoral closure using figure-of-eight stitch

INTERVENTIONS:
Procedure: Atrial Fibrillation with femoral closure using closing system — The ablation procedure will be performed under deep sedation/general anaesthesia as standard of care. Vital signs will be monitored. For patients on oral anticoagulation, the procedure will be performed according to the latest guidelines. For catheter access, sheaths will be placed in the femoral veins after ultrasound-guided puncture according to institutional standard. If the patient is randomised to the SDD group prior to the procedure, the femoral access will be closed with a closure system. Ablation technique, number of access points and procedural details will be performed according to institutional standard. Patients may be enrolled regardless of the energy source used for ablation. The minimum procedural endpoint is PVI. Ablation strategies in addition to PVI are at the discretion of the operator. Antiarrhythmic therapy may be administered for a maximum of 2 months (blanking period).
  Arms: SDD Group
Procedure: Atrial Fibrillation with femoral closure using figure-of-eight stitch — The ablation procedure will be performed under deep sedation/general anaesthesia as standard of care. Vital signs will be monitored. For patients on oral anticoagulation, the procedure will be performed according to the latest guidelines. For catheter access, sheaths will be placed in the femoral veins after ultrasound-guided puncture according to institutional standard. If the patient is randomised to the ONS group prior to the procedure, the femoral access will be closed with a figure-of-eight suture. The ablation technique, number of access points and procedural details will be performed according to institutional standard. Patients may be enrolled regardless of the energy source used for ablation. The minimum procedural endpoint is PVI. Ablation strategies in addition to PVI are at the discretion of the operator. Antiarrhythmic therapy may be administered for a maximum of 2 months (blanking period).
  Arms: ONS Group

SUMMARY:
Prospective, randomized, controlled, multicentre study to compare the safety and efficacy of a Same Day Discharge (SDD) protocol in combination with a Perclose ProStyle (PPS) /ProGlide (PPG) suture mediated vascular closure device to the current gold standard: an overnight stay (ONS) protocol associated with manual compression ± figure-of-eight suture for the patients receiving interventional pulmonary vein isolation (PVI).

DETAILED DESCRIPTION:
The aim of the study is to prove that the use of a SDD protocol does not lead to a higher rate of adverse events (minor and major), unplanned medical visits (emergency department or outpatients' clinic) and unplanned readmissions, while substantially reducing the costs associated with the medical care and increasing the comfort of the patients on a period of 30 days, when compared to ONS and manual compression ± figure-of-eight suture. Moreover, the safety, efficiency, and feasibility of the SDD protocol should be proven during a follow-up (FU) period of 12 months. The definition of endpoints will be trained in all participating study sites to preserve consistency.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >=18 years
* Elective catheter ablation for atrial fibrillation using 6 to 14 Fr inner diameter introducer sheath with a minimum of 1 and maximum of 2 femoral venous access sites, independent of the energy source use

Exclusion Criteria:

* Active systemic or cutaneous infection, or inflammation in vicinity of the groin
* Platelet count < 50,000 cells/mm3
* Body mass index (BMI) > 45 kg/m2 or < 18 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
30 Day vascular access-related adverse events | 30 days post intervention
  Primary Safety Endpoint
Time to ambulation | 2 Days after intervention
  Primary Efficacy Endpoint elapsed time between removal of the final closure device or removal of final sheath and the moment when the patient stood and walked 20 ft without evidence of venous re-bleeding from the femoral access site (time to ambulation; TTA)

SECONDARY OUTCOMES:
Quality of Life assessment - EQ-5D-5L | 12 Month after Intervention
  Secondary Efficacy Endpoint quality of life assessment (QoL) using the EQ-5D-5L questionnaire which contains 5 questions on current well-being and a scale from 0-100 on the personal assessment of the state of current health (from 0 (very poor) to 100 (very good)).
Quality of Life assessment - AFEQT | 12 Month after Intervention
  Secondary Efficacy Endpoint quality of life assessment (QoL) using the AFEQT questionnaire. which contains 20 questions on 7-point Likert scale on current well-being. Finally, a score between 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered) of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered)

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Tilz, Prof. Dr., Principal Investigator — Universitätsklinikum Schleswig-Holstein, Universitäres Herzzentrum Lübeck, Klinik für Rhythmologie; Sorin S Popescu, M.D., Study Chair — Universitätsklinikum Schleswig-Holstein, Universitäres Herzzentrum Lübeck, Klinik für Rhythmologie; Mirco Kuechler, M.Sc., Study Chair — Universitätsklinikum Schleswig-Holstein, Universitäres Herzzentrum Lübeck, Klinik für Rhythmologie, Studienzentrale
Locations (1):
- Klinik für Rhythmologie, Lübeck, Schleswig-Holstein, Germany